CLINICAL TRIAL: NCT02461186
Title: An Open-label Randomized Trial to Assess the Therapeutic Efficacy of Arterolane-piperaquine Versus Dihydroartemisinin-piperaquine for the Treatment of Uncomplicated Falciparum Malaria in Eastern Myanmar, an Area of Emerging Artemisinin-resistant Falciparum Malaria
Brief Title: Arterolane-PQP Versus DHA-PQP in Uncomplicated Falciparum Malaria in Eastern Myanmar
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Change of the study site due to the current political climate in Myanmar.
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); Department of Medical Research, Lower Myanmar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAKMAL1501
Record Dates: First submitted 2015-05-26; First posted 2015-06-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Uncomplicated Falciparum Malaria; Artemisinin-resistant
Keywords: Arterolane-piperaquine; Dehydroartemisinin-piperaquine; therapeutic efficacy; Uncomplicated falciparum malaria; Artemisinin-resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arterolane maleate-piperaquine phosphate (Synriam) (Experimental)
  Interventions: Drug: Arterolane maleate-piperaquine phosphate (Synriam)
- Dihydroartemisinin-piperaquine phosphate (Duocotexin) (Experimental)
  Interventions: Drug: Dihydroartemisinin-piperaquine phosphate (Duocotexin)

INTERVENTIONS:
Drug: Arterolane maleate-piperaquine phosphate (Synriam)
  Arms: Arterolane maleate-piperaquine phosphate (Synriam)
Drug: Dihydroartemisinin-piperaquine phosphate (Duocotexin)
  Arms: Dihydroartemisinin-piperaquine phosphate (Duocotexin)

SUMMARY:
Emerging resistance to artemisinins and their partner drugs severely threatens the treatment of falciparum malaria in Myanmar with artemisinin combination therapies. To inform drug policy, it is crucial to evaluate alternative antimalarial treatments.

The investigators here propose a randomized clinical trial comparing parasite clearance parameters and efficacy of 3 days arterolane-piperaquine with standard treatment with 3 days dihydroartemisinin (DHA)-piperaquine in adult patients with uncomplicated falciparum malaria in Myanmar stratified for the presence of "K13" mutation in the infecting parasite strains.

DETAILED DESCRIPTION:
Primary Objective:

- To assess the parasite clearance half-life of arterolane-piperaquine compared to DHA-piperaquine in patients with artemisinin resistant uncomplicated falciparum malaria, defined by presence of the "K13" mutations in the infecting parasite strain.

Secondary Objectives :

* To assess the therapeutic efficacy of arterolane-piperaquine and DHA-piperaquine for the treatment of uncomplicated falciparum malaria or mixed infection (P.falciparum (PF) + a non-falciparum species) at Day 42, stratified by presence of artemisinin resistance in the infecting parasite strain.
* To assess the frequency of adverse events and serious adverse events of arterolane-piperaquine compared to DHA-piperaquine.
* To assess other efficacy parameters related to parasite clearance and parasite cure rate as well as the gametocyte carriage.
* To obtain pharmacokinetic (PK) and pharmacokinetic/pharmacodynamics (PK/PD) data on arterolane-piperaquine and DHA-piperaquine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 year old
* Symptomatic malaria infection, i.e. history of fever or presence of fever >37.5°c (tympanic) within the last 24 hours.
* Microscopic confirmation of asexual stages of P.falciparum (may be mixed with non-falciparum species) with a parasitaemia >10,000 parasites/µL
* Able to take oral medication
* Willingness and ability of patients to comply with the study protocol for the duration of the study
* Written informed consent given to participate in the trial

Exclusion Criteria:

* Pregnancy or lactation (urine test for β HCG to be performed on any woman of child bearing age 18 to 45 year old)
* P.falciparum asexual stage parasitaemia greater than or equal to 4% red blood cells (175,000/µL).
* Signs or symptoms indicative of severe malaria:

  * Impaired consciousness
  * Severe anaemia (Hct<15%)
  * Bleeding disorder -evidenced by epistaxis, bleeding gums, frank haematuria, bleeding from venipuncture sites
  * Respiratory distress
  * Severe jaundice
* Have taken a full course DHA-piperaquine, artemether-lumefantrin or other antimalarial treatment in the previous 42 days
* Known hypersensitivity to artemisinins or to piperaquine - defined as history of erythroderma/other severe cutaneous reaction or angioedema
* History of splenectomy
* History of taking medicinal products that are known to prolong the QTc interval, including:

  * Antiarrhythmics (e.g. amiodarone, disopyramide, dofetilide, ibutilide, procainamide, quinidine, hydroquinidine, sotalol).
  * Neuroleptics (e.g. phenothiazines, sertindole, sultopride, chlorpromazine, haloperidol, mesoridazine, pimozide, or thioridazine), antidepressive agents.
  * Certain antimicrobial agents, including agents of the following classes:

    * macrolides (e.g. erythromycin, clarithromycin),
    * fluoroquinolones (e.g. moxifloxacin, sparfloxacin),
    * imidazole and triazole antifungal agent,
    * pentamidine and saquinavir.
  * The non-sedating antihistamines terfenadine, astemizole, mizolastine.
  * Other drugs: cisapride, droperidol, domperidone, bepridil, diphemanil, probucol, levomethadyl, methadone, vinca alkaloids, arsenic trioxide.
* History of taking any drug which is known to be metabolised by the cytochrome enzyme CYP2D6 including flecainide, metoprol, imipramine, amitriptyline, clomipramine.
* Family history of sudden unexplained death, or personal or family history of predisposing cardiac conditions for arrhythmia/QT prolongation (including congenital long QT syndrome, arrhythmia, QTc interval greater than 450 milliseconds with either Bazett or Fridericia correction).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Peripheral blood parasite half-life | 2 years
  Peripheral blood parasite half-life of the linear portion of the natural logarithm parasite clearance curve in patients with parasitaemia at inclusion >10,000 parasites/µL

SECONDARY OUTCOMES:
42 day PCR corrected adequate clinical and parasitological response (ACPR) | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Arjen M Dondorp, MD, Principal Investigator — Mahidol Oxfrod Tropical Medicine Research Unit